CLINICAL TRIAL: NCT06288984
Title: Effects of Repetitive Transcranial Magnetic Stimulation(rTMS) on Respiratory Function and Gut Microbiota in Patients With Brain Injury
Brief Title: Effects of rTMS on Respiratory Function and Gut Microbiota in Patients With Brain Injury
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NFEC-2024-061
Record Dates: First submitted 2024-02-17; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Brain Injuries; Respiratory Function Impaired; Gut Microbiota
MeSH Terms: conditions — Brain Injuries; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active rTMS (Experimental)
  Interventions: Device: active rTMS
- sham rTMS (Sham Comparator)
  Interventions: Device: sham rTMS

INTERVENTIONS:
Device: active rTMS — The magnetic stimulation coil was tangent to the scalp and kept parallel for 10 minutes a day, 5 days a week for 4 weeks
  Arms: active rTMS
Device: sham rTMS — The magnetic stimulation coil was tangent to the scalp and kept perpendicular for 10 minutes a day, 5 days a week for 4 weeks
  Arms: sham rTMS

SUMMARY:
Impaired respiratory function may occur after brain injury, and will progress to restricted respiratory dysfunction without early intervention. At present, there is a lack of effective treatment options for respiratory dysfunction. Repetitive Transcranial Magnetic Stimulation(rTMS) is a non-invasive, painless and non-invasive neuroregulatory technique. In healthy people, rTMS applied to the respiratory motor cortex induces a contralateral respiratory muscle response. However, whether rTMS can improve respiratory function in patients with brain injury remains unclear. gut microbiota can affect muscle function and mass, and animal experiments have shown that probiotics can increase skeletal muscle mass and grip strength in mice. On the other hand, studies have found that rTMS can improve the nutritional status of patients with vegetative state by regulating the structure of gut microbiota. However, it remains unclear whether rTMS can improve respiratory muscle function in patients with brain injury by regulating gut microbiota. Therefore, the investigators intend to apply rTMS to the respiratory motor cortex to observe whether rTMS can improve respiratory function and reduce the incidence of pneumonia in patients with brain injury, and to observe the role of gut microbiota in this process.

ELIGIBILITY:
Inclusion Criteria:

* In line with the diagnostic criteria of "Chinese classification of cerebrovascular diseases(2015)" mRS Score 2-4 points or craniocerebral injury caused by trauma, GCS score > 8 points
* Between 18 and 70 years old
* The first incidence of cerebrovascular disease or traumatic brain injury, and the course of disease was 10-180 days
* Vital signs are stable, no progression
* Voluntary participation with informed consent

Exclusion Criteria:

* Patients with a history of respiratory disease, including chronic bronchitis, chronic obstructive pulmonary disease, bronchiectasis, and lung cancer
* Severe bone malformations in the chest or spine
* Have other neurological or neuromuscular disorders
* History of thoracic and abdominal surgery
* Severe heart, lung, kidney, liver or other organ dysfunction
* Pregnant and lactating women
* Epilepsy
* Metal implant
* Patients who were judged by the investigator to be unsuitable for participation in this trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diaphragm thickness | Day 0，Week 4
  Diaphragm thickness was measured using a 10-15 MHz linear array probe, and the probe was positioned in the 8th to 11th costal space between the midaxillary line or anterior axillary line, perpendicular to the skin at the end of inspiratory phase and the end of expiratory phase.
Thickening fraction | Day 0，Week 4
  Thickening fraction = (end-inspiratory diaphragm thickness-end expiratory

SECONDARY OUTCOMES:
Diaphragm mobility | Day 0，Week 4
  Diaphragm mobility was measured with a 2-5MHz convex array probe, which was located below the costal arch of the midline of the clavicle. The above indexes were measured for 3 consecutive respiratory cycles and averaged.
Surface EMG of diaphragm | Day 0，Week 4
  The latency period, amplitude and motion threshold were determined by Transcranial magnetic stimulation of motor evoked potential(TMS-MEP).
Forced vital capacity(FVC) | Day 0，Week 4
  The FVC is measured using an Master-Screen spirometer
Forced expiratory volume at one second（FEV1） | Day 0，Week 4
  The FEV1 is measured using an Master-Screen spirometer
Peak expiratory flow (PEF) | Day 0，Week 4
  The PEF is measured using an Master-Screen spirometer
Maximum voluntary ventilation (MVV) | Day 0，Week 4
  The MVV is measured using an Master-Screen spirometer

IPD SHARING:
Plan to Share IPD: No